CLINICAL TRIAL: NCT06858865
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Safety and Pharmacokinetics of AD-228A Compared to Coadministration of AD-2281 and AD-2282 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of AD-228A Compared to Coadministration of AD-2281 and AD-2282
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-228BE-02
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Primary Hypercholesterolaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Experimental): Period 1 : Reference Drug(AD-2281 and AD-2282), Period 2 : Test Drug(AD-228A)
  Interventions: Drug: AD-228A; Drug: AD-2281 and AD-2282
- Sequence B (Experimental): Period 1 : Test Drug(AD-228A), Period 2 : Reference Drug(AD-2281 and AD-2282)
  Interventions: Drug: AD-228A; Drug: AD-2281 and AD-2282

INTERVENTIONS:
Drug: AD-228A — AD-228A Oral Tablet
Drug: AD-2281 and AD-2282 — AD-2281 Oral Tablet + AD-2282 Oral Tablet

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-228A in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety profiles of AD-228A compared with coadministration AD-2281 and AD-2282 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose to 72 hours
  Cmax of AD-228A
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose to 72 hours
  AUCt of AD-228A

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No